CLINICAL TRIAL: NCT06134440
Title: ImmunoNutrition and Colorectal Adenocarcinoma Surgery: a Randomized Study. INCAS Study
Brief Title: ImmunoNutrition and Colorectal Adenocarcinoma Surgery - INCAS Study
Acronym: INCAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOV-CRC-01-2022 INCAS
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, open-label, single-centre study in patients candidate to elective curative surgery for colon-rectal cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (interventional arm) (Experimental): a low-fiber dietary advice + oral nutritional supplement enriched with immune-nutrients for 5 pre-operative days and 5 post-operative days.
  Interventions: Dietary Supplement: Impact Oral®
- Arm B (control arm) (No Intervention): a low fiber dietary advice only

INTERVENTIONS:
Dietary Supplement: Impact Oral® — All patients will follow low-fiber diet according to ERAS protocol during the study period. Patients assigned to the experimental arm will assume also Impact Oral®, an oral nutritional supplement with immune-nutrients (hyper-proteic formula), manufactured and commercialized by Nestlé Health Science S.p.a. It is a liquid drink packaged in a brick of 237 ml. Patients will assume Impact Oral® for 5 days before surgery and 5 day after surgery.
  Arms: Arm A (interventional arm)

SUMMARY:
Compared to upper gastrointestinal (GI) malignancies, CRC patients generally present with satisfactory nutritional status at surgery and malnutrition is typically present in advanced stages of CRC. Therefore, in the latter surgery may not be offered with curative intent. Based on the current evidence, the role of OIN appears to be consolidated for malnourished patients undergoing surgery for gastrointestinal cancer. Regarding not malnourished patients, there is still no clear correlation between OIN and decrease in post-operative complications. Furthermore, whether OIN increases immune response within the tumour microenvironment is based on studies with poor number of patients.

DETAILED DESCRIPTION:
Randomized, controlled, open-label, single-centre study in patients candidate for elective curative surgery for colon-rectal cancer.

The study intervention consists of the oral nutritional supplementation enriched with immune-nutrients delivered before and after surgery in addition to standard dietary advice according to E.R.A.S. protocol.

All patients will follow low-fiber diet according to ERAS protocol during the study period. Patients assigned to the experimental arm will assume also Impact Oral®, an oral nutritional supplement with immune-nutrients (hyper-proteic formula), manufactured and commercialized by Nestlé Health Science S.p.a. It is a liquid drink packaged in a brick of 237 ml. Patients will assume Impact Oral® for 5 days before surgery and 5 day after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years or older;
* histologically confirmed adenocarcinoma of colon or rectum;
* Eligible for elective curative surgery with indication of colon and/or rectal resection in laparoscopy with mini-invasive technique;
* eligible for ERAS protocol;
* Written informed consent to the study participation according to the Local Ethic Committee requirements before any study procedure;

Exclusion Criteria:

* colon or rectal resection for benign disease;
* TNM Stage ≥4;
* neoadjuvant radio and/or chemotherapy
* ASA score > 3;
* contraindications to oral nutrition (e.g. dysphagia, pyloric stenosis) or hypersensitivity to any ingredient of study product;
* albuminemia < 3.0 g/l;
* weight loss > 10% in the last 3-6 months;
* BMI < 18.5 kg/m2;
* pregnant or breastfeeding;
* Not self-sufficient or with poor family compliance;
* Congenital or acquired immunodeficiency;
* Active uncontrolled pre-operative infections or other clinically relevant concomitant illness that preclude laparoscopic procedure;
* Bowel obstruction or parenteral nutrition or gastric tube;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure - Number of patients with grade 2 or higher post-operative complications | within 30 days post-surgical intervention
  Number of patients with grade 2 or higher post-operative complications according to Clavien-Dindo classification occurred within 30 days post-surgical intervention.

SECONDARY OUTCOMES:
Secondary Outcome Measure - Hospital length of stay | From the day of surgery until discharge, assessed up to 7 days
  Hospital length of stay defined as hospitalization from the day of surgery until discharge
Secondary Outcome Measure - Reoperation rate | within 30 days following the index surgery
  Reoperation rate within 30 days from index surgery defined as any unplanned post-operative procedure including a return in the operating room or an imaging-guided intervention within 30 days following the index surgery
Secondary Outcome Measure - Unplanned readmissions | within 30 days from discharge
  Unplanned readmissions within 30 days from discharge
Secondary Outcome Measure - 30-day mortality for any cause | 30-day mortality for any cause
  30-day mortality for any cause
Secondary Outcome Measure - Safety assessed according to CTCAE | From admission to discharge, assessed up to 42 days
  Safety assessed according to criteria to NCI Common Toxicity Criteria Adverse Event (CTCAE), version 5
Secondary Outcome Measure - Nutritional status before and after surgery | differences at day 1, 3, 5, 15 and 30 after surgery from T0 (7-10 days before surgery) will be calculated and compared between the two arms
  Nutritional status before and after surgery will be assessed evaluating albumin, prealbumin and transferrin serum levels: differences at day 1, 3, 5, 15 and 30 after surgery from T0 (7-10 days before surgery) will be calculated and compared between the two arms
Secondary Outcome Measure - Inflammatory status before and after surgery | differences at day 1, 3, 5, 15 and 30 after surgery from T0 (7-10 days before surgery) will be calculated and compared between the two arms
  Inflammatory status before and after surgery will be assessed evaluating leukocytes (x10^(9)/L), C-reactive protein (PCR) (mg/dL), procalcitonin (ug/L), neutrophil-lymphocyte (ratio), and lactate dehydrogenase (LDH) serum levels (U/L).
  The haematic quantification of this biomarkers provides information about the inflammatory status.

OTHER OUTCOMES:
Translational Outcome Measures - Evaluation of the immune-modulatory effects of OIN in the tumor micro-environment in CRC patients | The analysis will be performed 7 days before surgery and 5 days after surgery.
  To evaluate the immune-modulatory effects of OIN in the tumor micro-environment in CRC patients. Immunological assessment of adaptive and innate immune cells will be investigated on pre-operative biopsy and surgical specimen by immunohistochemistry (IHC), and pre and post-treatment on peripheral blood by flow cytometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Oncologico Veneto IRCCS, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided